CLINICAL TRIAL: NCT01192867
Title: A Phase III, Multi-Center, Randomized, 24 Week, Double-Blind, Parallel-Group, Placebo-Controlled Study to Evaluate Efficacy and Safety of RO4917838 in Stable Patients With Persistent, Predominant Negative Symptoms of Schizophrenia Treated With Antipsychotics Followed by a 28 Week, Double-Blind Treatment Period
Brief Title: A Study of RO4917838 in Participants With Persistent, Predominant Negative Symptoms of Schizophrenia (NN25310)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN25310; 2010-020370-42 (EudraCT Number)
Record Dates: First submitted 2010-08-30; First posted 2010-09-01 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- RO4917838 20 milligrams (mg) (Experimental): Participants, on stable antipsychotics, will receive RO4917838 orally at 20 mg once daily (QD) up to 56 weeks followed by an optional treatment extension for up to 3 years.
  Interventions: Drug: RO4917838; Drug: Antipshychotics (Standard of Care)
- RO4917838 10 mg (Experimental): Participants, on stable antipsychotics, will receive RO4917838 orally at 10 mg QD up to 56 weeks followed by an optional treatment extension for up to 3 years.
  Interventions: Drug: RO4917838; Drug: Antipshychotics (Standard of Care)
- Placebo (Placebo Comparator): Participants, on stable antipsychotics, will receive RO4917838 matching placebo orally QD up to 56 weeks.
  Interventions: Drug: Placebo; Drug: Antipshychotics (Standard of Care)

INTERVENTIONS:
Drug: Placebo — Placebo will be administered orally QD for 56 weeks
  Arms: Placebo
Drug: RO4917838 — RO4917838 will be administered orally at 20 or 10 mg QD for 56 weeks.
  Arms: RO4917838 10 mg; RO4917838 20 milligrams (mg)
Drug: Antipshychotics (Standard of Care) — Participants will continue to receive their stable antipshychotic as standard of care based on their prescription up to Week 56.

SUMMARY:
This multi-center, randomized, double-blind, parallel-group, placebo-controlled study will evaluate the efficacy and safety of RO4917838 in participants with persistent, predominant negative symptoms of schizophrenia. Participants, on stable treatment with antipsychotics, will be randomized to receive daily oral doses of RO4917838 or matching placebo for 56 weeks (treatment period 1 of 24 weeks and treatment period 2 of 32 weeks), followed by an optional treatment extension for up to 3 years. After 52 weeks, participants who were originally randomized to an active treatment will be randomly assigned to receive either placebo or continue on the originally assigned study treatment for 4 weeks washout period (Week 52 to Week 56) for the assessment of potential withdrawal effects in a blinded manner using participants staying on active treatment as a control. Participants initially randomized to placebo will remain on placebo. After 56 weeks, participants who were switched to placebo in the washout period will return to their blinded, active treatment arm.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia of paranoid, disorganized, residual, undifferentiated or catatonic subtype
* Predominant negative symptoms
* With the exception of clozapine, participants are on any of the available marketed atypical or typical antipsychotics (treatment with a maximum of two antipsychotics)

Exclusion Criteria:

* Evidence that participant has clinically significant, uncontrolled and unstable disorder (e.g. cardiovascular, renal, hepatic disorder)
* Body Mass Index (BMI) of less than (<) 17 or greater than (>) 40 kilograms per meter square (kg/m^2)
* Depressive symptoms, defined as a score of 9 or greater on the Calgary Depression Rating Scale for Schizophrenia (CDSS)
* A severity score of 3 or greater on the Parkinsonism item of the Exrapyramidal Symptoms Rating Scale-Abbreviated (ESRS-A) (Clinical Global Impression, Parkinsonism)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 629 (Actual)
Dates: Start 2010-12-11 (Actual); Primary Completion 2014-05-26 (Actual); Study Completion 2014-05-26 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in the Positive and Negative Symptoms Scales (PANSS) Negative Symptoms Factor Score at Week 24 (All-Participant Population) | Baseline, Week 24
Percentage of Participants With Adverse Events (All-Participant Population) | Week 24

SECONDARY OUTCOMES:
Change From Baseline in the PANSS Negative Symptoms Factor Score at Week 24 (Complement Factor H Related Protein 1 High [CFHR1-High] Subgroup Population) | Baseline, Week 24
Change From Baseline in the Personal and Social Performance (PSP) Total Score at Week 24 (All-Participant Population) | Baseline, Week 24
Change From Baseline in the PSP Total Score at Week 24 (CFHR1-High Subgroup Population) | Baseline, Week 24
Change From Baseline in the PANSS Total Score at Week 24 (All-Participant Population) | Baseline, Week 24
Change From Baseline in the PANSS Total Score at Week 24 (CFHR1-High Subgroup Population) | Baseline, Week 24
Change From Baseline in the PANSS Factor Score at Week 24 (All-Participant Population) | Baseline, Week 24
Change From Baseline in the PANSS Factor Score at Week 24 (CFHR1-High Subgroup Population) | Baseline, Week 24
Change From Baseline in the PANSS Subscale Scores at Week 24 (All-Participant Population) | Baseline, Week 24
Change From Baseline in the PANSS Subscale Scores at Week 24 (CFHR1-High Subgroup Population) | Baseline, Week 24
Percentage of Participants Who Have at least 20 Percent (%) Improvement From Baseline in the PANSS Negative Symptom Factor Score at Week 24 (All-Participant Population) | Baseline, Week 24
Percentage of Participants Who Have at least 20% Improvement From Baseline in the PANSS Negative Symptom Factor Score at Week 24 (CFHR1-High Subgroup Population) | Baseline, Week 24
Percentage of Participants Who Have at least 20% Improvement From Baseline in the PANSS Negative Symptom Factor Score for Two out of Three Assessments During 24 Weeks (All-Participant Population) | Baseline up to Week 24
Percentage of Participants Who Have at least 20% Improvement From Baseline in the PANSS Negative Symptom Factor Score for Two out of Three Assessments During 24 Weeks (CFHR1-High Subgroup Population) | Baseline up to Week 24
Percentage of Participants With Improvement From Baseline in the Overall Clinical Status Based on Clinical Global Impression - Improvement (CGI-I) Score (All-Participant Population) | Baseline, Week 24
Percentage of Participants With Improvement From Baseline in the Overall Clinical Status Based on CGI-I Score (CFHR1 Subgroup Population) | Baseline, Week 24
Percentage of Participants With Improvement From Baseline in the Overall Clinical Status Based on CGI-I Score for Two out of Three Assessments During 24 Weeks (All-Participant Population) | Baseline up to Week 24
Percentage of Participants With Improvement From Baseline in the Overall Clinical Status Based on CGI-I Score for Two out of Three Assessments During 24 Weeks (CFHR1 Subgroup Population) | Baseline up to Week 24
Percentage of Participants With Improvement From Baseline in the Negative Symptoms Based on CGI-I Negative Symptoms Score (All-Participant Population) | Baseline, Week 24
Percentage of Participants With Improvement From Baseline in the Negative Symptoms Based on CGI-I Negative Symptoms Score (CFHR1 Subgroup Population) | Baseline, Week 24
Percentage of Participants With Improvement From Baseline in the Negative Symptoms Based on CGI-I Negative Symptoms Score for Two out of Three Assessments During 24 Weeks (All-Participant Population) | Baseline up to Week 24
Percentage of Participants With Improvement From Baseline in the Negative Symptoms Based on CGI-I Negative Symptoms Score for Two out of Three Assessments During 24 Weeks (CFHR1 Subgroup Population) | Baseline up to Week 24
Percentage of Participants Who Have at least 20% Improvement From Baseline in the PANSS Negative Symptom Factor Score at Week 24 and Improvement in the Negative Symptoms Based on CGI-I Negative Symptoms Score (All-Participant Population) | Baseline, Week 24
Percentage of Participants Who Have at least 20% Improvement From Baseline in the PANSS Negative Symptom Factor Score at Week 24 and Improvement in the Negative Symptoms Based on CGI-I Negative Symptoms Score (CFHR1 Subgroup Population) | Baseline, Week 24
Change From Baseline in Severity of Illness Based on Clinical Global Impression - Severity (CGI-S) Overall Score (All-Participant Population) | Baseline, Week 24
Change From Baseline in Severity of Illness Based on CGI-S Overall Score (CFHR1 Subgroup Population) | Baseline, Week 24
Change From Baseline in Severity of Illness Based on CGI-S Negative Symptoms Score (All-Participant Population) | Baseline, Week 24
Change From Baseline in Severity of Illness Based on CGI-S Negative Symptoms Score (CFHR1 Subgroup Population) | Baseline, Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (122):
- United States (27):
  - K&S Professional Research Services LLC, Little Rock, Arkansas
  - Advanced Research Center Inc., Anaheim, California
  - Comprehensive Clinical Development- Cerritos CA, Cerritos, California
  - Diligent Clinical Trials Inc, Downey, California
  - Care Research Center, La Palma, California
  - Pasadena Research Institute, Pasadena, California
  - CNRI - Los Angeles, LLC, Pico Rivera, California
  - Pharmax Research Clinic Inc., Miami, Florida
  - Northwest Behavioral Research Center, Marietta, Georgia
  - American Medical Research, Inc, Oak Brook, Illinois
  - University of Iowa College of Medicine; Psychiatry Research, Iowa City, Iowa
  - Clinical Insights, Inc., Glen Burnie, Maryland
  - St Louis Clinical Trials, St Louis, Missouri
  - Ocean Rheumatology, Toms River, New Jersey
  - CRI Worldwide LLC, Willingboro, New Jersey
  - Raymond G. Murphy VA Medical Center, Albuquerque, New Mexico
  - Behavioral Medical Research of Brooklyn, Brooklyn, New York
  - Comprehensive NeuroScience, Fresh Meadows, New York
  - North Carolina Psychiatric Research Center, Raleigh, North Carolina
  - UC Health Clinical Trials Office, Cincinnati, Ohio
  - Belmont Center for Comprehensive Treatment; Research, Philadelphia, Pennsylvania
  - Claghorn-Lesem Research Clinic, Inc., Bellaire, Texas
  - FutureSearch Clinical Trials, LP, Dallas, Texas
  - Pillar Clinical Research LLC, Dallas, Texas
  - Family Psychiatry of the Woodlands P.A., The Woodlands, Texas
  - Pacific Institute of Medical Sciences, Bothell, Washington
  - Eastside Therapeutic Resource, Kirkland, Washington
- Argentina (13):
  - Centro SERES, Buenos Aires
  - Fundacion para el Estudio y Tratamiento des las Enfi Mentales, Buenos Aires
  - Mulieris, CABA
  - Facene Fund.Argentina Contra Enferm.Neur.Del Envejecimiento, Ciudad Autonoma Bs As
  - Instituto Nacional de Psicopatologia, Ciudad Autonoma Bs As
  - Instituto DAMIC - Fundación Rusculleda, Córdoba
  - Sanatorio Prof.Leon.S.Morra S.A, Córdoba
  - Instituto de Neurociencias San Agustín S.A., La Plata
  - Centro de Psiquiatria Biologica Professor Julio J. Herrera; Psiquiatria, Mendoza
  - Resolution Psicopharmacology Research Institute, Mendoza
  - Centro de Asistencia e Investigación en Neurociencias, Mendoza
  - CIAP - Centro de Investigacion y Asistencia en Psiquiatria, Rosario
  - Centro de Investigacion Clinica Farmacologica en Psiquiatria, Santiago del Estero
- Australia (4):
  - Westmead Hospital; Department of Psychiatry, Westmead, New South Wales
  - Monash Medical Centre-Clayton Campus; School of Psychology and Psychiatry, Clayton, Victoria
  - Frankston Hospital; Mental Health Service, Frankston, Victoria
  - The Alfred Hospital; Monash Alfred Psychiatry Research Centre (MAP-RC), Melbourne, Victoria
- Colombia (3):
  - Centro de Investigaciones y Proyectos en Neurociencias CIPNA, Barranquilla
  - E.S.E. Hospital Mental de Antioquia, Bello
  - Centro de Investigaciones del Sistema Nervioso Limitada - Gr, Bogotá
- Privater, Kuopio, Finland
- France (7):
  - Centre Hospitalier Universitaire Caen; Pôle Psychiatrie - Addictologie, Caen
  - CHU Gabriel Montpied; Service de Psychiatrie, Clermont-Ferrand
  - Centre Hospitalier Specialise du Jura, Dole
  - Cabinet Médical Ambroise Paré, Élancourt
  - Hôpital de la Conception; Pôle Psychiatrique Centre, Marseille
  - CHU Strasbourg Nouvel Hôpital Civil;Service de Psychiatrie I, Strasbourg
  - Hopital Chalucet; Unite de Psychiatrie, Toulon
- Hungary (8):
  - Dr. Kenessey Albert Hospital; Psychiatry I., Balassagyarmat
  - Fov.Onk.Szt Janos Korh. E-Budai Egyesitett Korhazai; Pszichiatriaci rehabilitacio, Budapest
  - Semmelweis Egyetem AOK; Pszichiatriai es Pszichoterapias Klinika, Budapest
  - Fovarosi Onkormanyzat Nyiro Gyula Korhaza; Pszichatria II, Budapest
  - Fovarosi Onkormanyzat Nyiro Gyula Korhaza; Pszichiatria I., Budapest
  - UNO Medical Trials Kft., Budapest
  - Petz Aladar Megyei Oktato Korhaz; Pszichiatria I., Győr
  - Békés Megyei Pándy Kálmán Kórház; Onkologiai tanszek, Gyula
- India (10):
  - Samvedna Hospitals; Samvedana Psychiatry and Sex Therapy Hospital, Ahmedabad
  - Sneh Clinic, Ahmedabad
  - Gujarat Institute of Psychological Research (GIPS), Ahmedabad
  - Mental Health Care & Research, Jaipur
  - R. K.Yadav Memorial Mental Health & De-Addiction Hospital, Jaipur
  - Manav Neuropsychiatric Hospital Pvt. Ltd., Kalyān
  - Kasturba Medical College & Hospital, Mangalore
  - K. S. Hegde Medical Academy, Mangalore
  - Poona Hospital and Research Centre, Pune
  - Brij Psychiatry Hospital & Muskaan Research Centre; Maanav Health Foundation, Vadodara
- Mexico (5):
  - Arete Proycectos y Administracion S.C, México
  - Centro de Investigacion Medica S.C; Hospital Santa Cecilia de Monterrey S.A. de C.V., Monterrey
  - Medikalink, Monterrey
  - Instituto de informacion e investigacion en salud mental AC, Monterrey
  - Hospital Lomas de San Luis Internacional, San Luis Potosí City
- Romania (10):
  - Spitalul Clinic Judetean Arad; Departamentul de Psihiatrie, Arad
  - Spit Univ Urgenta Militar Dr. Carol Davila; Sectia Psihiatrie, Bucharest
  - Spitalul Clinic de Psihiatrie Prof. Dr. Alexandru Obregia; Clinical III Psihiatrie, Bucharest
  - Spitalul Clinic de Psihiatrie Prof. Dr. Alexandru Obregia; Comunitara si Reintegrare Psihosociala, Bucharest
  - Spitalul Clinic de Psihiatrie Prof. Dr. Alexandru Obregia; Sectia Clinica XIII Psihiatrie, Bucharest
  - Spitalul Clinic Judetean de Urgenta Cluj; Sectia Clinica de Psihiatrie III, Cluj-Napoca
  - Spitalul Universitar de Psihiatrie Socola, Lasi
  - Spitalul Clinic Municipal Dr. Gavril Curteanu; Sectia Clinica Psihiatrie I, Oradea
  - Spitalul de Psihiatrie Dr. Gh. Preda Sibiu;CSM Adulti Sibiu, Sibiu
  - Cabinet Medical S.C. Lorentina 2102 S.R.L.; Psihiatrie, Targouiste
- Russia (18):
  - Kemerovo Regional Clinical Psychiatric Hospital, Kemerovo
  - GUZ Lipetsk Regional psychoneurological Hospital #1; Dispansary Department, Lipetsk
  - Scientifically Research Institute of Psychiatry of Ministry of Health of the Russian Federation, Moscow
  - Institution of RAMS (Mental Health Research Center of RAMS), Moscow
  - Federal State Institution Moscow SRI of Psychiatry of Minzdravsocrazvitia, Moscow
  - Central Moscow Regional Clinical Psychiatric Hospital, Moscow
  - Moscow Region Psychiatric Hospital #5, Moscow Region
  - City Clinical Psychiatry Hospital #1, Nizhny Novgorod
  - St. Petersburg State Healthcare Institution, Saint Petersburg
  - City Psychiatric Hospital #2 of St. Nikolay Chudotvorets, Saint Petersburg
  - Saint Petersburg Psychoneurological Research Institute of Roszdrav n.a. Bekhterev, Saint Petersburg
  - St. Petersburg GUZ City Psychiatric Hospital #6, Saint Petersburg
  - Military Medical Academy, Saint Petersburg
  - St. Petersburg State Healthcare Institution "City Mental Hospital #3; I.I. Skvortsov-Stepanov, Saint Petersburg
  - Samara Psychiatric Hospital, Samara
  - Mhi City Clinical Hospital #2 Named After v.i. Razumousky, Sartatov
  - Arkhangelsk Regional Clinical Psychiatric Hospital, Talagi
  - Tomsk Clinical Psychiatric Hospital, Tomsk
- South Korea (9):
  - Inje University Busan Paik Hospital, Busan
  - Chonnam National University Hospital, Gwangju
  - Korea University Ansan Hospital, Gyeonggi-do
  - Inha University Hospital, Incheon
  - Gil Hospital. Gachon University, Incheon
  - Chonbuk National Uni Hospital, Jeollabuk-do
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - The Catholic University of Korea St.Mary's Hospital, Seoul
- Sweden (4):
  - Integrerad Närsjukvård i Malmö, Malmo
  - Karolinska Universitetssjukhuset Huddinge, Psykiatri Sydväst, Stockholm
  - Danderyds Sjukhus AB; PRIMA Vuxenpsykiatri, Stockholm
  - Akademiska Sjukhuset; Psykosvård och rättspsykiatrisk vård, Uppsala
- United Kingdom (3):
  - Royal Edinburgh Hospital; Psychiatry, Edinburgh
  - Institute of Pyschiatry, London
  - Wareneford Hospital, Oxford

REFERENCES:
- [Derived] Georgiades A, Davis VG, Atkins AS, Khan A, Walker TW, Loebel A, Haig G, Hilt DC, Dunayevich E, Umbricht D, Sand M, Keefe RSE. Psychometric characteristics of the MATRICS Consensus Cognitive Battery in a large pooled cohort of stable schizophrenia patients. Schizophr Res. 2017 Dec;190:172-179. doi: 10.1016/j.schres.2017.03.040. Epub 2017 Apr 20. PMID 28433500
- [Derived] Bugarski-Kirola D, Blaettler T, Arango C, Fleischhacker WW, Garibaldi G, Wang A, Dixon M, Bressan RA, Nasrallah H, Lawrie S, Napieralski J, Ochi-Lohmann T, Reid C, Marder SR. Bitopertin in Negative Symptoms of Schizophrenia-Results From the Phase III FlashLyte and DayLyte Studies. Biol Psychiatry. 2017 Jul 1;82(1):8-16. doi: 10.1016/j.biopsych.2016.11.014. Epub 2016 Dec 15. PMID 28117049